CLINICAL TRIAL: NCT01981681
Title: A Phase 1, Randomized, Third-Party Open, Placebo-Controlled, Multiple Dose Escalation, Parallel Group Study To Evaluate Local Tolerability, Safety And Pharmacokinetics Of Topically Applied PF-06263276 In Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate Tolerability, Safety, And Pharmacokinetics Of Topical PF-06263276 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B5391002; 2013-004231-68
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Placebo-Controlled; Multiple Dose Escalation; Tolerability; Safety; PK; Topical; Healthy; PF-06263276

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 Experimental Arm (Experimental)
  Interventions: Drug: PF-06263726
- Cohort 2 Experimental Arm (Experimental)
  Interventions: Drug: PF-06263726
- Cohort 3 Experimental Arm (Experimental)
  Interventions: Drug: PF-06263726
- Cohort 3 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 4 Experimental Arm (Experimental)
  Interventions: Drug: PF-06263726
- Cohort 4 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06263726 — Subjects will receive dose strength of 2% PF-06263276 (1.14 mg) and matching placebo in topical formulation (2.5 µL/cm2) to be applied twice daily to two separate contralateral 20 cm2 areas on the back.
  Arms: Cohort 1 Experimental Arm
Drug: PF-06263726 — Subjects will receive dose strength of 4% PF-06263276 (2.28 mg) and matching placebo in topical formulation (2.5 µL/cm2) to be applied twice daily to two separate contralateral 20 cm2 areas on the back.
  Arms: Cohort 2 Experimental Arm
Drug: PF-06263726 — Subjects will receive dose strength of 2% PF-06263276 (11.4 mg) in topical formulation (2.5 µL/cm2) to be applied twice daily to a 200 cm2 area on the back.
  Arms: Cohort 3 Experimental Arm
Drug: Placebo — Subjects will receive dose strength of 2% PF-06263276 (11.4 mg) matching placebo in topical formulation (2.5 µL/cm2) to be applied twice daily to a 200 cm2 area on the back.
  Arms: Cohort 3 Placebo Arm
Drug: PF-06263726 — Subjects will receive dose strength of 4% PF-06263276 (22.8 mg) in topical formulation (2.5 µL/cm2) to be applied twice daily to a 200 cm2 area on the back.
  Arms: Cohort 4 Experimental Arm
Drug: Placebo — Subjects will receive dose strength of 4% PF-06263276 (22.8 mg) matching placebo in topical formulation (2.5 µL/cm2) to be applied twice daily to a 200 cm2 area on the back.
  Arms: Cohort 4 Placebo Arm

SUMMARY:
PF-06263276 is a first in class inhibitor of the Janus kinase (JAK) enzymes 1, 2, 3 and tyrosine kinase 2 (TYK2) that is being developed for the treatment of chronic plaque psoriasis. The goal of the study is to assess the safety, local tolerability, and pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects willing to avoid tanning beds and sun exposure of the back during the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of application).
* Subjects with any active skin condition at the application site possibly affecting drug absorption (e.g. rash, sun burn, scars, tattoos).
* Subjects with a Draize score >0 of the test area (back) immediately prior to first treatment application.
* Subjects using topical prescription or nonprescription drugs/over the counter preparations on the back within 14 days of the first treatment application.
* Subjects not willing to avoid application of treatmentssuch as lotions or creams to the back throughout the study until follow-up.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Draize toxicity assessment score. | Day 8, Day 28
  Changes from baseline on Draize toxicity assessment score.
Changes from baseline vital signs (blood pressure, pulse rate, oral temperature and respiration rate) and physical examinations. | Day 23, Day 28
Changes from baseline in 12 lead electrocardiogram (ECG) parameters. | Day 23, Day 28
  Quantitative changes in ECG intervals.
Incidence and severity of treatment emergent adverse events and withdrawals due to treatment emergent adverse events. | Day 23, Day 28
Incidence and magnitude of treatment emergent clinical laboratory abnormalities including hematology, chemistry, fasting glucose, urinalysis. | Day 23, Day 28

SECONDARY OUTCOMES:
Cohorts 3 and 4: Maximum Observed Plasma Concentration (Cmax) | Day 1, Day 14
Cohorts 3 and 4: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1, Day 14
Cohorts 3 and 4: Area Under the Curve From Time Zero to 12 hours [AUC (0-12)] | Day 1, Day 14
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Cohorts 3 and 4: Dose-Normalized Area Under the Curve From Time Zero to 12 hours [AUC (0-12)] | Day 1, Day 14
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Cohorts 3 and 4: Dose-Normalized Maximum Observed Plasma Concentration [Cmax (dn)] | Day 1, Day 14
Cohorts 3 and 4: Plasma Decay Half-Life (t1/2) | Day 14
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Cohorts 3 and 4: Apparent Volume of Distribution (Vz/F) | Day 14
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Cohorts 3 and 4: Apparent Oral Clearance (CL/F) | Day 14
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5391002&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20Tolerability%2C%20Safety%2C%20And%20Pharmacokinetics%20Of%20Topical%20PF-06263276%20In%20Healthy%20Subjects